CLINICAL TRIAL: NCT06045468
Title: Observational Study on Early Rehabilitation After Transfemoral Amputation in Moderately Active Patients, Provided With Kenevo (Ottobock)
Brief Title: Early Rehabilitation After Transfemoral Amputation in Moderately Active Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Median (Other)
Collaborators: Otto Bock Healthcare Products GmbH (Industry); University Medical Center Mainz (Other)
Responsible Party: Principal Investigator, Johannes Schroeter, Director of Orthopaedic clinic, Median
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Kenevo2023
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Transfemoral Amputation
Keywords: Kenevo; MPK; specialized inpatient rehabilitation

STUDY DESIGN:
Intervention Model Description: Non-randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients in inpatient rehabilitation in study center.
  Interventions: Other: Amputation-specialized rehabilitation
- Control group (Experimental): Patients in inpatient rehabilitation facility of collaborating clinics.
  Interventions: Other: Non-amputation-specialized rehabilitation

INTERVENTIONS:
Other: Amputation-specialized rehabilitation — Study center; amputation-specialized unit within rehabilitation facility; fully practicing national guidelines
  Arms: Study group
Other: Non-amputation-specialized rehabilitation — Control clinics; treating some amputated patients each year but do not practice national guidelines or partially practicing national guidelines
  Arms: Control group

SUMMARY:
Treatment and rehabilitation after transfemoral amputation represents a challenging medical field, involving intersectoral parties. Although treatment guidelines exists, their implementation is difficult. This study is conducted to evaluate the need to practice these guidelines in order to gain best benefits for the patients. Focus is set of early inpatient rehabilitation and the role of a microprocessor-controlled prothesis (Kenevo, Ottobock).

DETAILED DESCRIPTION:
Right after major surgeries, e.g. amputations, inpatient rehabilitation follows in Germany. Costs are covered by different insurances, like public or private health care insurances or German pension insurance. Usually, inpatient rehabilitation lasts for 3 weeks. But after some surgeries, like amputation, patients need more time to recover and fitting of a prosthesis takes additional time. Therefore guidelines state, that rehabilitation should take up to 6-8 weeks after major amputation. To provide evidence to these guidelines, we conducted this study.

Patients' choice on rehabilitation clinic decides on their assignment to the study group or control group. Inpatient rehabilitation is monitored with outcomes measurements. 3 measurements are carried out in the study group within rehabilitational stay of around 6 weeks (admission - middle - discharge) and 2 measurements are carried out in the control group within rehabilitational stay of around 3 weeks (admission - discharge). After discharge from rehabilitation, assessment of patient reported outcome measurements is continued every 6 weeks for both groups. Follow-up phase ends with 24 weeks after admission to rehabilitation.

For subanalysis, different prosthetic devices (non-microprocessor-controlled vs. microprocessor-controlled prosthesis) are compared.

ELIGIBILITY:
Inclusion Criteria:

* inpatient rehabilitation stay after transfemoral amputation or knee disarticulation
* anticipated K-level 1 or 2
* body weight no more than 125kg (authorized body weight for prosthetic device)
* German speaking
* able to give informed consent

Exclusion Criteria:

* non-German speaking
* not able to give informed consent
* body weight over 125kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Limb User's Survey of Mobility (PLUS-M) | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  Patient reported outcome measurement with 12 questions assessing mobility; reported as t-score, max. t-score: 65.7

SECONDARY OUTCOMES:
Reintegration to normal living index (RNLI) | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  Patient reported outcome measurement with 11 questions asking to patients' reintegration into daily life, reported as percentage
EuroQol questionnaire (EQ-5D-5L) | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  Patient reported outcome measurement assessing quality of life, reported as health utility, score, score 0-1 with 0 meaning lowest quality of life and 1 highest quality of life
Falls | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  Number of falls with prothesis
Fear of falling | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  indoor and outdoor fear of falling on a numeric rating scale (0-10) with 0 meaning no fear of falling and 10 meaning maximum fear of falling
Locomotor capability index (LCI 5) | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  Patient reported outcome measurement assessing patients' locomotor capability, 14 questions, results are categorized in 2 dimension: basic or advanced activities, maximum score is 28 points for each dimension
Barthel Index | As follow-up 24 weeks after admission to rehabilitation (around 18-21 weeks after discharge from rehabilitation)
  Patient reported outcome measurement assessing patients' self care, 10 questions with maximum score of 100 points
Timed Up and Go Test | At admission to rehabilitation facility (if patients are already equipped with a prosthesis), after 3 weeks and after 6 weeks (discharge from rehabilitation) of inpatient rehabilitation stay
  Functional outcome measurement, assessing patients' capability to walk, time needed to get up from a chair, walk 3 m, turn and walk 3 m back until sitting down again
6 minute walking test | At admission to rehabilitation facility (if patients are already equipped with a prosthesis), after 3 weeks and after 6 weeks (discharge from rehabilitation) of inpatient rehabilitation stay
  Patient walks back and forth 12 m for 6 minutes, distance in meter is recorded
AMP-PRO | At admission to rehabilitation facility (if patients are already equipped with a prosthesis), after 3 weeks and after 6 weeks (discharge from rehabilitation) of inpatient rehabilitation stay
  Functional outcome measurement, amputated-specific, assesses different activities of daily life, max. score 43 points

CONTACTS AND LOCATIONS:
Locations (1):
- MEDIAN Clinics, Wiesbaden, Germany